CLINICAL TRIAL: NCT00655863
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing SYR-322 Alone and Combination SYR-322 With Pioglitazone Versus Placebo on Postprandial Lipids in Subjects With Type 2 Diabetes
Brief Title: Efficacy of Alogliptin and With Pioglitazone in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322_301; 2007-000486-38 (EudraCT Number); U1111-1113-2081 (Registry Identifier: WHO); NL22649.029.08 (Registry Identifier: CCMO)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg QD + Pioglitazone 30 mg QD (Experimental)
  Interventions: Drug: Alogliptin and Pioglitazone

INTERVENTIONS:
Drug: Alogliptin and Pioglitazone — Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 16 weeks.
  Other Names: alogliptin; SYR110322; Actos; AD-4833; SYR-322
  Arms: Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 16 weeks.
  Other Names: SYR110322; SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Placebo — Alogliptin placebo-matching tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 16 weeks.
  Other Names: Actos; AD-4833; SYR-322
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to compare the efficacy of Alogliptin, once daily (QD), taken by itself and with pioglitazone on postprandial lipid measures in type 2 diabetes.

DETAILED DESCRIPTION:
SYR-322 (alogliptin) is a selective, orally available inhibitor of dipeptidyl peptidase IV being developed as a treatment for type 2 diabetes mellitus. Dipeptidyl peptidase IV is the primary enzyme involved in the in vivo degradation of at least 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide.

Pioglitazone HCl (ACTOS®) is a thiazolidinedione developed by Takeda Chemical Industries, Ltd. (Osaka, Japan). Pioglitazone HCl depends on the presence of insulin for its mechanism of action.

This study will assess the effects of alogliptin and alogliptin coadministered with pioglitazone HCl on postprandial lipid and lipoprotein metabolism in participants with type 2 diabetes. Individuals who participate in this study will be required to commit to a screening visit and up to 6 additional visits at the study center. Study participation is anticipated to be about 20 weeks (or approximately 5 months). Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations and electrocardiograms. At 3 of the visits a meal will be served that must be eaten within 10 minutes.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of type 2 diabetes
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Either failed treatment with diet and exercise for 3 months prior to Screening or has been receiving a stable dose of metformin, sulfonylurea, nateglinide, or repaglinide for more than 3 months prior to Screening.
* Inadequate glycemic control as defined by glycosylated hemoglobin concentration between 6.5 and 9.0%, inclusive.
* Fasting plasma glucose less than 13.3 mmol per L.
* Fasting serum triglyceride level of 1.7 to 5.0 mmol per L, inclusive.
* Has not been receiving any lipid-lowering therapy within 3 months prior to Screening or on a stable statin and/or ezetimibe therapy (same drug and dose) for at least 3 months.
* Body mass index greater than 23 kg/m2 and less than 45 kg/m2.
* If has regular use of other, non-excluded medications, must be on a stable dose for at least 4 weeks prior to Screening. Use of as needed prescription medications and over-the-counter medications is allowed at the discretion of the investigator.
* Is to be Apolipoprotein E 3/3 or Apolipoprotein E 3/4 phenotype positive prior to baseline.

Exclusion Criteria

* History of type 1 diabetes.
* History of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years.
* Diastolic blood pressure greater than 100 mm Hg or a systolic blood pressure of greater than 160 mm Hg.
* History of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study medication.
* Hemoglobin less than 120 g per L for males and less than100 g per L for females.
* Alanine transaminase level greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
* Serum creatinine level greater than 133 μmol per L.
* Fasting total cholesterol greater than 6.5 mmol per L.
* New York Heart Association heart failure of any Class (I-IV) regardless of therapy.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within 6 months prior to Screening.
* History of acute metabolic diabetic complications.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with human immunodeficiency virus.
* History of diabetic gastro paresis.
* History of gastric bypass surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- Amsterdam, Netherlands
- Gothenburg, Sweden

REFERENCES:
- [Result] Eliasson B, Moller-Goede D, Eeg-Olofsson K, Wilson C, Cederholm J, Fleck P, Diamant M, Taskinen MR, Smith U. Lowering of postprandial lipids in individuals with type 2 diabetes treated with alogliptin and/or pioglitazone: a randomised double-blind placebo-controlled study. Diabetologia. 2012 Apr;55(4):915-25. doi: 10.1007/s00125-011-2447-3. Epub 2012 Jan 12. PMID 22237690
- See also: ACTOS Package Insert. — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 2 investigative sites in The Netherlands and Sweden from 16 July 2007 to 17 December 2009.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Placebo QD: Alogliptin placebo-matching tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 16 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 16 weeks.
- Alogliptin 25 mg QD + Pioglitazone 30 mg QD: Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 16 weeks.
Period: Overall Study
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Started | 24 | 25 | 22
Completed | 24 | 25 | 21
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD | Total
Number analyzed (Participants) | 24 | 25 | 22 | 71
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (6.23) | 58.7 (6.47) | 59.1 (6.94) | 59.0 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 7 | 21
  Male | 20 | 15 | 15 | 50
Region of Enrollment [Number; unit: participants]
  Netherlands | 9 | 10 | 9 | 28
  Sweden | 15 | 15 | 13 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants] — White
  Participants | 24 | 25 | 22 | 71
Weight [Mean (Standard Deviation); unit: kg] | 101.83 (11.989) | 93.68 (10.816) | 93.05 (13.160) | 96.24 (12.471)
Height [Mean (Standard Deviation); unit: cm] | 178.3 (6.74) | 173.9 (8.17) | 172.8 (10.97) | 175.0 (8.91)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.12 (3.997) | 31.09 (4.196) | 31.15 (3.503) | 31.46 (3.898)
Diabetes duration [Mean (Standard Deviation); unit: years] | 5.55 (3.243) | 6.40 (3.622) | 5.03 (3.791) | 5.69 (3.548)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Postprandial Incremental Area Under the Curve for Total Triglycerides at Week 16.
Description: The change in postprandial (after eating a meal) incremental area under the plasma concentration-time curve from 0 to 8 hours (AUC (0-8h)) postdose at week 16 relative to baseline.
Time Frame: Baseline and Week 16.
Population: The full analysis set included all randomized participants who took at least 1 dose of double-blind study medication. Participants who were in the full analysis set and had a baseline and at least 1 post-baseline assessment were included for this analysis. Missing values were imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mg.h/dL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 21
mg.h/dL | -39.728 (48.2481) | -346.957 (47.2251) | -293.439 (51.1271)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 25 mg QD; The null hypothesis that there was no difference between Alogliptin 25 mg QD and placebo groups was tested at a 2-sided 0.05 significance level. The ANCOVA model used for the change in postprandial incremental area the curver for total triglycerides includes treatment and statin use as fixed effects and baseline AUC(0-8h) for total triglycerides as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value and confidence interval presented without multiplicity adjustment; Mean Difference (Final Values) = -307.229, 95% CI 2-sided [-443.168 to -171.290]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD + Pioglitazone 30 mg QD; The null hypothesis that there was no difference between Alogliptin 25 mg QD + Pioglitazone 30 mg QD and placebo QD groups was tested at a 2-sided 0.05 significance level. The ANCOVA model used for the change in postprandial incremental area the curve for total triglycerides includes treatment and statin use as fixed effects and baseline AUC(0-8h) for total triglycerides as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value and confidence interval presented without multiplicity adjustment; Mean Difference (Final Values) = -253.711, 95% CI [-394.161 to -113.262]

2. Secondary Outcome: Change From Baseline in Postprandial Incremental Area Under the Curve for Total Triglycerides at Week 4.
Description: The change in postprandial incremental area under the plasma concentration-time curve from 0 to 8 hours (AUC(0-8h)) postdose at week 4 relative to baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg.h/dL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 21 | 19
mg.h/dL | -16.291 (61.1286) | -288.490 (65.4530) | -279.116 (68.4947)

3. Secondary Outcome: Change From Baseline in Postprandial Incremental Area Under the Curve Changes for Lipid Parameters.
Description: The change in postprandial incremental area under the plasma concentration-time curve for very-low-density lipoprotein (VLDL) cholesterol, VLDL triglycerides, VLDL2 cholesterol, VLDL2 triglycerides, chylomicron cholesterol, chylomicron triglycerides, intermediate-density lipoprotein (IDL) cholesterol, and IDL triglycerides from 0 to 8 hours postdose at week 4 and week 16 relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg.h/dL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
mg.h/dL
  VLDL triglycerides Week 4 (n=23; n=21; n=19) | -9.488 (35.4108) | -119.009 (37.0255) | -98.758 (38.9818)
  VLDL triglycerides Week 16 (n=23; n=25; n=21) | 25.194 (29.4896) | -130.459 (28.2397) | -85.709 (30.7867)
  VLDL cholesterol Week 4 (n=23; n=21; n=19) | -6.914 (4.3110) | -14.760 (4.4843) | -10.760 (4.7065)
  VLDL cholesterol Week 16 (n=23; n=25; n=21) | -4.561 (3.4790) | -16.365 (3.3125) | -8.747 (3.5984)
  VLDL 2 triglycerides Week 4 (n=23; n=20; n=19) | -5.221 (7.8102) | -17.960 (8.3710) | -8.687 (8.6678)
  VLDL 2 triglycerides Week 16 (n=23; n=25; n=21) | -24.280 (3.4497) | -18.986 (3.3104) | -23.061 (3.6369)
  VLDL 2 cholesterol Week 4 (n=23; n=20; n=19) | -2.396 (0.8474) | -0.709 (0.9059) | -1.073 (0.9345)
  VLDL 2 cholesterol Week 16 (n=23; n=25; n=21) | -2.190 (0.7833) | -1.445 (0.7506) | -1.232 (0.8217)
  Chylomicron triglycerides Week 4 (n=23; n=21; n=1 | 0.617 (26.1603) | -115.093 (27.4280) | -108.036 (28.6857)
  Chylomicron triglycerides Week 16(n=23;n=25; n=21) | -18.577 (15.2943) | -136.626 (14.6683) | -129.991 (15.9053)
  Chylomicron cholesterol Week 4 (n=23; n=21; n=19) | -0.091 (1.1845) | -4.474 (1.2425) | -3.628 (1.3039)
  Chylomicron cholesterol Week 16 (n=23; n=25; n=21) | -1.431 (0.6001) | -5.566 (0.5769) | -4.289 (0.6265)
  IDL triglycerides Week 4 (n=22; n=18; n=17) | 14.667 (12.9991) | -6.771 (14.3964) | -4.410 (14.9182)
  IDL triglycerides Week 16 (n=22; n=23; n=19) | -0.313 (2.9265) | -4.045 (2.8759) | -4.533 (3.1885)
  IDL cholesterol Week 4 (n=22; n=18; n=17) | 1.473 (1.5215) | -0.808 (1.6835) | 0.195 (1.7328)
  IDL cholesterol Week 16 (n=22; n=23; n=19) | 0.171 (0.6006) | 0.249 (0.5893) | 0.609 (0.6499)

4. Secondary Outcome: Change From Baseline in Postprandial Incremental Area Under the Curve for Lipoprotein Parameters.
Description: Postprandial incremental area under the curve changes for very-low-density lipoprotein (VLDL) Apo B-48, VLDL Apo B 100, VLDL2 Apo B-48, VLDL2 Apo B 100, chylomicron Apo B-48, chylomicron Apo B 100, and intermediate density lipoprotein (IDL) Apo B-48, IDL Apo B 100, and triglyceride-rich remnant (TRR) lipoproteins from 0 to 8 hours postdose at week 4 and week 16 relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg.h/dL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
mg.h/dL
  VLDL apo B-48 Week 4 (n=19; n=12; n=15) | -0.020 (0.2902) | -0.491 (0.3572) | -0.312 (0.3180)
  VLDL apo B-48 Week 16 (n=19; n=16; n=16) | -0.055 (0.1956) | -0.654 (0.2077) | -0.266 (0.2044)
  VLDL apo B 100 Week 4 (n=19; n=12; n=15) | 0.568 (2.2981) | -2.670 (2.8906) | -2.977 (2.5811)
  VLDL apo B 100 Week 16 (n=19; n=16; n=16) | -0.453 (1.8388) | -6.967 (2.0109) | -3.265 (2.0025)
  VLDL2 apo B-48 Week 4 (n=19; n=12; n=15) | -0.075 (0.0776) | -0.101 (0.0969) | -0.022 (0.0870)
  VLDL2 apo B-48 Week 16 (n=19; n=16; n=16) | -0.079 (0.0674) | -0.175 (0.0732) | 0.002 (0.0737)
  VLDL2 apo B 100 Week 4 (n=19; n=12; n=15) | 0.464 (1.1846) | 0.507 (1.4982) | -0.781 (1.33287)
  VLDL2 apo B 100 Week 16 (n=19; n=16; n=16) | -1.155 (0.7985) | -2.049 (0.8732) | -1.793 (0.8707)
  Chylomicron apo B-48 Week 4 (n=19; n=12; n=14) | -0.051 (0.0236) | -0.097 (0.0302) | -0.071 (0.0272)
  Chylomicron apo B-48 Week 16 (n=19; n=16; n=16) | -0.051 (0.0180) | -0.113 (0.0197) | -0.084 (0.0191)
  Chylomicron apo B 100 Week 4(n=19; n=12; n=14) | -0.123 (0.0825) | -0.417 (0.1041) | -0.389 (0.0960)
  Chylomicron apo B 100 Week 16 (n=19; n=16; n=16) | -0.120 (0.0544) | -0.419 (0.0594) | -0.409 (0.0590)
  IDL apo B-48 Week 4 (n=18; n=10; n=13) | 0.002 (0.1254) | -0.247 (0.1707) | -0.223 (0.1476)
  IDL apo B-48 Week 16 (n=18; n=14; n=14) | 0.151 (0.1368) | -0.188 (0.1580) | 0.021 (0.1561)
  IDL apo B 100 Week 4 (n=18; n=10; n=13) | 0.952 (3.3778) | -2.029 (4.5494) | -2.769 (3.8565)
  IDL apo B 100 Week 16 (n=18; n=14; n=14) | 4.181 (3.4923) | -2.876 (3.9944) | 0.073 (3.8906)
  TRR lipoproteins Week 4 (n=24; n=21; n=19) | 16.147 (5.6739) | -1.071 (6.0930) | -5.673 (6.4428)
  TRR lipoproteins Week 16 (n=24; n=25; n=21) | 2.818 (3.1250) | -12.719 (3.0884) | -7.853 (3.3658)

5. Secondary Outcome: Postprandial Changes Over Time From Baseline for Glucagon-like Peptide-1 (GLP-1)
Description: Postprandial changes over time at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
pmol/L
  Week 4: 1 hour postprandial (n=20; n=17; n=15) | 0.52 (1.167) | -5.48 (1.249) | -4.88 (1.330)
  Week 4: 2 hours postprandial (n=21; n=17; n=16) | 0.92 (1.524) | -2.93 (1.702) | -6.41 (1.732)
  Week 4: 3 hours postprandial (n=21; n=17; n=16) | 1.20 (1.619) | -2.08 (1.789) | -3.61 (1.848)
  Week 4: 4 hours postprandial (n=21; n=17; n=16) | 1.76 (1.823) | 2.86 (2.027) | -0.84 (2.077)
  Week 4: 8 hours postprandial (n=19; n=16; n=16) | -1.01 (0.955) | -0.38 (1.039) | -0.72 (1.040)
  Week 16: 1 hour postprandial (n=21 ; n=20; n=16) | -0.28 (1.304) | -4.10 (1.326) | -3.63 (1.462)
  Week 16: 2 hours postprandial (n=21; n=21; n=17) | -3.59 (1.451) | -3.75 (1.457) | -3.75 (1.599)
  Week 16: 3 hours postprandial (n=21; n=21; n=17) | -1.08 (1.206) | -2.25 (1.202) | -3.17 (1.326)
  Week 16: 4 hours postprandial (n=21; n=21; n=17) | -0.64 (1.263) | -1.88 (1.271) | -1.83 (1.393)
  Week 16: 8 hours postprandial (n=21; n=21; n=17) | -1.36 (0.820) | 0.03 (0.819) | -1.48 (0.910)

6. Secondary Outcome: Postprandial Changes Over Time From Baseline for Glucose
Description: Postprandial changes over time at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
mg/dL
  Week 4: 1 hour postprandial (n=24; n=21; n=19) | -5.957 (5.3970) | -35.065 (5.7617) | -65.905 (6.0315)
  Week 4: 2 hours postprandial (n=23; n=21; n=19) | -4.049 (5.9932) | -24.721 (6.2299) | -67.718 (6.5647)
  Week 4: 3 hours postprandial (n=24; n=21; n=18) | 3.200 (6.3047) | -19.367 (6.7356) | -54.345 (7.2106)
  Week 4: 4 hours postprandial (n=24; n=21; n=19) | 2.930 (5.3775) | -13.907 (5.6699) | -48.643 (6.0151)
  Week 4: 8 hours postprandial (n=22; n=21; n=19) | 0.046 (4.1120) | -6.077 (4.2043) | -27.856 (4.3961)
  Week 16: 1 hour postprandial (n=24; n=25; n=21) | 11.867 (8.1356) | -36.189 (7.9793) | -58.168 (8.6585)
  Week 16: 2 hours postprandial (n=23; n=25; n=21) | 17.324 (8.6572) | -29.745 (8.2830) | -61.899 (9.0248)
  Week 16: 3 hours postprandial (n=24; n=25; n=20) | 18.379 (7.8017) | -16.996 (7.6465) | -51.891 (8.4838)
  Week 16: 4 hours postprandial (n=24; n=25; n=21) | 10.849 (7.3084) | -12.517 (7.1054) | -41.943 (7.7396)
  Week 16: 8 hours postprandial (n=24; n=25; n=21) | 3.266 (5.0112) | -5.737 (4.9335) | -19.381 (5.3350)

7. Secondary Outcome: Postprandial Changes Over Time From Baseline for Insulin
Description: Postprandial changes over time at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
uIU/mL
  Week 4: 1 hour postprandial (n=24; n=21; n=18) | -5.047 (3.5562) | -5.867 (3.7749) | -18.287 (4.0906)
  Week 4: 2 hours postprandial (n=24; n=21; n=19) | 1.405 (6.3051) | 3.161 (6.7294) | -28.700 (7.0572)
  Week 4: 3 hours postprandial (n=24; n=21; n=19) | 0.637 (5.2789) | 0.652 (5.6125) | -18.842 (5.9301)
  Week 4: 4 hours postprandial (n=24; n=21; n=19) | 2.999 (3.5652) | 5.092 (3.8075) | -12.891 (4.0088)
  Week 4: 8 hours postprandial (n=23; n=21; n=19) | -1.174 (1.0270) | 2.685 (1.0772) | -6.000 (1.1301)
  Week 16: 1 hour postprandial (n=24; n=25; n=21) | -8.896 (4.8993) | -14.368 (4.7784) | -12.162 (5.2052)
  Week 16: 2 hours postprandial (n=24; n=25; n=21) | -9.258 (6.5119) | -9.528 (6.4000) | -24.777 (6.9371)
  Week 16: 3 hours postprandial (n=24; n=25; n=21) | 4.447 (4.8889) | -9.848 (4.7800) | -23.025 (5.2049)
  Week 16: 4 hours postprandial (n=24; n=25; n=21) | 8.405 (4.5090) | -4.753 (4.4158) | -19.329 (4.8159)
  Week 16: 8 hours postprandial (n=24; n=25; n=21) | 0.495 (1.2847) | 3.163 (1.2637) | -6.107 (1.3728)

8. Secondary Outcome: Postprandial Changes Over Time From Baseline for Glucagon
Description: Postprandial changes over time at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
pg/mL
  Week 4: 1 hour postprandial (n=24; n=21; n=19) | 7.222 (3.7636) | -14.639 (4.0619) | -17.704 (4.2418)
  Week 4: 2 hours postprandial (n=24; n=21; n=19) | 1.730 (3.3262) | -17.015 (3.5627) | -22.081 (3.7541)
  Week 4: 3 hours postprandial (n=24; n=21; n=19) | 6.637 (3.7141) | -13.200 (3.9753) | -15.987 (4.2015)
  Week 4: 4 hours postprandial (n=24; n=20; n=18) | 2.021 (4.1496) | -4.679 (4.5627) | -8.860 (4.7910)
  Week 4: 8 hours postprandial (n=22; n=20; n=19) | 1.081 (3.5000) | -3.789 (3.6665) | -5.150 (3.7592)
  Week 16: 1 hour postprandial (n=24; n=25; n=21) | 3.318 (3.1819) | -16.955 (3.1477) | -17.462 (3.4144)
  Week 16: 2 hours postprandial (n=24; n=25; n=21) | -1.047 (3.4159) | -20.949 (3.3556) | -20.662 (3.6653)
  Week 16: 3 hours postprandial (n=24; n=25; n=21) | 4.842 (3.4670) | -13.602 (3.4048) | 10.84 (3.7260)
  Week 16: 4 hours postprandial (n=24; n=24; n=21) | 2.801 (3.1830) | -8.577 (3.1873) | -10.326 (3.4011)
  Week 16: 8 hours postprandial (n=24; n=25; n=21) | 3.917 (2.5383) | -5.818 (2.4876) | -9.332 (2.7108)

9. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 8 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 21
percentage of glycosylated hemoglobin
  Week 8: fasting (n=23; n=24; n=20) | -0.12 (0.084) | -0.55 (0.083) | -1.01 (0.090)
  Week 16: 5 minutes prior to meal (n=24;n=25; n=21) | 0.38 (0.131) | -0.39 (0.129) | -0.95 (0.140)

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change in fasting plasma glucose collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4, Week 8 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
mg/dL
  Week 4 (n=24; n=20; n=19) | -4.141 (3.0027) | -20.669 (3.3024) | -38.826 (3.3890)
  Week 8 (n=24; n=25; n=21) | 4.864 (5.3254) | -16.293 (5.2451) | -38.242 (5.7203)
  Week 16 (n=24; n=25; n=21) | 11.869 (6.4897) | -17.052 (6.3918) | -38.481 (6.9709)

11. Secondary Outcome: Change From Baseline in Postprandial C-Peptide
Description: The change in postprandial C-peptide collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
ng/mL
  Week 4: 1 hour postprandial (n=24; n=21; n=19) | -0.106 (0.2597) | -0.300 (0.2775) | -1.199 (0.2921)
  Week 4: 2 hours postprandial (n=24; n=21; n=19) | 0.311 (0.3789) | -0.011 (0.4052) | -1.379 (0.4262)
  Week 4: 3 hours postprandial (n=24; n=21; n=19) | 0.376 (0.4386) | 0.116 (0.4684) | -1.230 (0.4933)
  Week 4: 4 hours postprandial (n=24; n=21; n=19) | 0.256 (0.3674) | 0.393 (0.3926) | -1.173 (0.4140)
  Week 4: 8 hours postprandial (n=23; n=20; n=19) | -0.063 (0.1530) | 0.421 (0.1643) | -0.911 (0.1699)
  Week 16: 1 hour postprandial (n=24; n=25; n=21) | -0.176 (0.3474) | -1.021 (0.3405) | -0.646 (0.3712)
  Week 16: 2 hours postprandial (n=24; n=25; n=21) | -0.011 (0.4337) | -1.006 (0.4259) | -1.055 (0.4638)
  Week 16: 3 hours postprandial (n=24; n=25; n=21) | 0.492 (0.4570) | -0.712 (0.4478) | -1.269 (0.4882)
  Week 16: 4 hours postprandial (n=24; n=25; n=21) | 0.496 (0.4042) | -0.068 (0.3961) | -1.515 (0.4323)
  Week 16: 8 hours postprandial (n=24; n=24; n=21) | 0.151 (0.2042) | 0.588 (0.2047) | -0.761 (0.2194)

12. Secondary Outcome: Change From Baseline in Postprandial Proinsulin
Description: The change in postprandial proinsulin collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
pmol/L
  Week 4: 1 hour postprandial (n=24; n=21; n=19) | -4.555 (3.9248) | -13.024 (4.2068) | -41.192 (4.4562)
  Week 4: 2 hours postprandial (n=24; n=21; n=19) | -0.208 (5.5216) | -12.568 (5.9505) | -56.478 (6.3185)
  Week 4: 3 hours postprandial (n=24; n=21; n=19) | -6.735 (5.9547) | -12.987 (6.4485) | -59.573 (6.8034)
  Week 4: 4 hours postprandial (n=24; n=21; n=19) | -6.496 (5.9756) | -6.848 (6.4875) | -52.649 (6.8526)
  Week 4: 8 hours postprandial (n=23; n=21; n=19) | -5.082 (4.3735) | -5.561 (4.6395) | -35.159 (4.9287)
  Week 16: 1 hour postprandial (n=24; n=25; n=21) | 2.081 (5.3253) | -22.812 (5.2274) | -30.658 (5.7287)
  Week 16: 2 hours postprandial (n=24; n=25; n=21) | 3.336 (6.3373) | -29.930 (6.2396) | -45.487 (6.8516)
  Week 16: 3 hours postprandial (n=24; n=25; n=21) | 5.863 (6.2769) | -27.768 (6.2041) | -50.058 (6.7783)
  Week 16: 4 hours postprandial (n=24; n=25; n=21) | 8.671 (5.7153) | -21.862 (5.6549) | -48.757 (6.1834)
  Week 16: 8 hours postprandial (n=24; n=25; n=21) | 6.935 (5.2859) | -6.898 (5.2307) | -28.776 (5.7372)

13. Secondary Outcome: Change From Baseline in High-sensitive C-reactive Protein (Hs-CRP)
Description: The change in hs-CRP collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
mg/L
  Week 4: 5 minutes prior to meal (n=24; n=21; n=19) | -1.514 (1.0846) | 0.631 (1.1693) | 0.155 (1.2269)
  Week 16: 5 minutes prior to meal (n=24; n=25;n=21) | 4.338 (2.6070) | -0.402 (2.5683) | -0.402 (2.8000)

14. Secondary Outcome: Change From Baseline in Adiponectin
Description: The change in adiponectin collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 21
µg/mL
  Week 4: 5 minutes prior to meal (n=24;n=21; n=19) | 0.001 (0.0004) | 0.000 (0.0005) | 0.006 (0.0005)
  Week 16: 5 minutes prior to meal (n=24;n=25;n=21) | 0.000 (0.0005) | 0.000 (0.0005) | 0.007 (0.0005)

15. Secondary Outcome: Change From Baseline in Anti-Vascular Cell Adhesion Molecule (VCAM)
Description: The change in VCAM collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 21
ng/mL
  Week 4: 5 minutes prior to meal (n=24;n=21; n=19) | -37.351 (17.6828) | 2.392 (18.8767) | 4.849 (19.8297)
  Week 16: 5 minutes prior to meal (n=24;n=25;n=21) | 5.067 (16.6654) | -1.441 (16.3094) | 13.665 (17.7580)

16. Secondary Outcome: Change From Baseline in Anti-Intercellular Adhesion Molecule (ICAM)
Description: The change in ICAM collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 21
ng/mL
  Week 4: 5 minutes prior to meal (n=24;n=21; n=19) | -1.154 (6.7415) | -0.294 (7.1785) | -23.810 (7.6380)
  Week 16: 5 minutes prior to meal (n=24; n=25;n=21) | -2.495 (8.6653) | -4.140 (8.4752) | -16.556 (9.3414)

17. Secondary Outcome: Change From Baseline in e-Selectin
Description: The change in e-Selectin collected at each week indicated relative to baseline.
Time Frame: Baseline, Week 4 and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
ng/mL
  Week 4: 5 minutes prior to meal (n=24;n=21; n=19) | 1.041 (1.3484) | 0.116 (1.4394) | -6.437 (1.5137)
  Week 16: 5 minutes prior to meal (n=24; n=25;n=21) | 1.488 (2.0944) | -1.671 (2.0480) | -4.056 (2.2336)

18. Secondary Outcome: Change From Baseline in Endothelial Function Through Pulse Wave Tonometry
Description: Pulse wave tonometry performed before the meal and 2 hours postmeal using one recording consisting of 15 to 20 sequentially recorded radial artery waveforms collected at each assessment.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Number analyzed (Participants) | 24 | 25 | 22
mmHg
  Week 16: pre-meal (n=23;n=23;n=20) | -3.6 (2.51) | -4.7 (2.52) | -4.2 (2.68)
  Week 16: 2 hours postmeal (n=24;n=24;n=20) | -1.6 (3.16) | 0.1 (3.18) | -1.3 (3.47)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory values or ECG findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo QD | Alogliptin 25 mg QD | Alogliptin 25 mg QD + Pioglitazone 30 mg QD
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/25 | 3/22
Other Adverse Events (participants affected / at risk) | 15/24 | 19/25 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=24) | Alogliptin 25 mg QD (N=25) | Alogliptin 25 mg QD + Pioglitazone 30 mg QD (N=22)
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=24) | Alogliptin 25 mg QD (N=25) | Alogliptin 25 mg QD + Pioglitazone 30 mg QD (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 5 | 3
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.